CLINICAL TRIAL: NCT06323356
Title: A Phase 3, Open-Label, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of TAK-279 in Adult Subjects With Generalized Pustular Psoriasis or Erythrodermic Psoriasis
Brief Title: A Study of TAK-279 in Adult Participants With Generalized Pustular Psoriasis or Erythrodermic Psoriasis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-279-PsO-3005; jRCT2031230714 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Generalized Pustular Psoriasis; Erythrodermic Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAK-279 for Generalized Pustular Psoriasis (Experimental): Participants with generalized pustular psoriasis will receive TAK-279 from Day 1 up to Week 52.
  Interventions: Drug: TAK-279
- TAK-279 for Erythrodermic Psoriasis (Experimental): Participants with erythrodermic psoriasis will receive TAK-279 from Day 1 up to Week 52.
  Interventions: Drug: TAK-279

INTERVENTIONS:
Drug: TAK-279 — Specified drug on specified days.

SUMMARY:
The main aim of this study is to check if TAK-279 improves symptoms of With Generalized Pustular Psoriasis (GPP) or Erythrodermic Psoriasis (EP) and side effect from the study treatment or TAK-279.

All participants will be assigned to study treatments of TAK-279 and will be treated with TAK-279 if the participants meet the study rules.

Participants will be in the study for up to 61 weeks including 52 weeks of study treatment. During the study, participants will visit their study clinic for multiple times.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of GPP or EP prior to the screening visit.
2. Candidate for phototherapy or systemic therapy.

Exclusion Criteria:

1. Other forms of psoriasis.
2. History of recent infection.
3. Any prior exposure to TAK-279, or participation in any study that included a TYK2 inhibitor.

Other protocol defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Static Physician's Global Assessment (sPGA) of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Week 16 | Baseline, Week 16
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving ≥75% Improvement from Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 16 | Baseline, Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.

SECONDARY OUTCOMES:
Percentage of Participants Achieving an sPGA of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Week 52 | Baseline, Week 52
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving an sPGA of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Both Week 16 and Week 52 Visits | Baseline, Week 16 and Week 52
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving an sPGA of Clear (0) at Week 16 and Week 52 | Week 16 and Week 52
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' will include all participants who score a 0.
Percentage of Participants Achieving an sPGA of Clear (0) or Almost Clear (1) at Week 16 and Week 52 | Week 16 and Week 52
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving an sPGA of Clear (0) or Almost Clear (1) at Week 16 and Week 52 Visits | Week 16 and Week 52
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving PASI-75 at Week 52 | Week 52
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-90 at Week 16 and Week 52 | Week 16 and Week 52
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 90% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-100 at Week 16 and Week 52 | Week 16 and Week 52
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing 100% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-75 at Both the Week 16 and Week 52 Visits | Week 16 and Week 52
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score at both the Week 16 and Week 52 visits relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-90 at Both the Week 16 and Week 52 Visits | Week 16 and Week 52
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 90% improvement in PASI score at both the Week 16 and Week 52 visits relative to baseline PASI score will be reported.
Percentage of Participants Achieving a Scalp-specific Physician's Global Assessment (ssPGA) of Absence of Disease (0) or Very Mild Disease (1) With a ≥2-Point Decrease from Baseline at Week 16 and Week 52 | Week 16 and Week 52
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate worsening.
Change from baseline in ssPGA at Weeks 16 and 52 | Baseline, Week 16 and Week 52
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate worsening.
Percentage of Participants Achieving a PGA of the Hands and/or Feet of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Weeks 16 and Week 52 | Baseline, Week 16 and Week 52
  PGA is a 5-point scale and a score of 0 to 4 should be assigned, based on the category that best describes the severity of active psoriasis of the participant's hands and feet, where 0=clear and 4=severe. Higher scores indicate worsening of severity. It will be evaluated for participants with the presence of active hand or foot psoriasis on Day 1.
Percentage of Participants with a Baseline Dermatology Life Quality Index (DLQI) Score ≥2 who Achieve DLQI Score of 0 or 1 at Week 16 and Week 52 | Week 16 and Week 52
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's quality of life (QoL) during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life).
Change from Baseline in DLQI at Week 16 and Week 52 | Baseline, Week 16 and Week 52
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life).
Change from Baseline in Nail Psoriasis Severity Index (NAPSI) at Week 16 and Week 52 Among Participants with Nail Involvement at Baseline | Baseline, Week 16 and Week 52
  The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lunula, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each nail will be scored for both nail matrix and nail bed psoriasis for each quadrant (ranging from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores indicate more severe psoriasis.
Change from Baseline in Body Surface Area (BSA) Affected by Psoriasis at Week 16 and Week 52 | Baseline, Week 16 and Week 52
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement.
Percentage of Participants with Generalized Pustular Psoriasis Who Achieve a Generalized Pustular Psoriasis Global Assessment (GPPGA) Pustulation Subscore of No Visible Pustules (0) at Week 16 and Week 52 | Week 16 and Week 52
  GPPGA is common endpoints in clinical studies of Generalized Pustular Psoriasis (GPP), and is skin-based scoring systems. The GPPGA is a clinician assessment of overall GPP severity based on a modified PGA, and the severity of pustules, erythema, and scaling of GPP lesions will be assessed. The five grades of severity for erythema, scaling, and pustulation correspond to 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. The GPPGA score is based on averaging the individual scores for erythema, scaling, and pustulation ranging from 0 to 4. Higher scores indicate more severe GPP.
Percentage of Participants with Generalized Pustular Psoriasis Who Achieve a GPPGA of Clear (0) or Almost Clear (1) at Weeks 16 and Week 52 | Week 16 and Week 52
  GPPGA is common endpoints in clinical studies of Generalized Pustular Psoriasis (GPP), and is skin-based scoring systems. The GPPGA is a clinician assessment of overall GPP severity based on a modified PGA, and the severity of pustules, erythema, and scaling of GPP lesions will be assessed. The five grades of severity for erythema, scaling, and pustulation correspond to 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. The GPPGA score is based on averaging the individual scores for erythema, scaling, and pustulation ranging from 0 to 4. Higher scores indicate more severe GPP.
Percentage of Participants with Generalized Pustular Psoriasis Who Achieve a GPPGA of Clear (0) at Week 16 and Week 52 | Week 16 and Week 52
  GPPGA is common endpoints in clinical studies of Generalized Pustular Psoriasis (GPP), and is skin-based scoring systems. The GPPGA is a clinician assessment of overall GPP severity based on a modified PGA, and the severity of pustules, erythema, and scaling of GPP lesions will be assessed. The five grades of severity for erythema, scaling, and pustulation correspond to 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. The GPPGA score is based on averaging the individual scores for erythema, scaling, and pustulation ranging from 0 to 4. Higher scores indicate more severe GPP.
Percentage of Participants with Generalized Pustular Psoriasis Who Achieve ≥75% Improvement from Baseline in Generalized Pustular Psoriasis Area and Severity Index (GPPASI) Score at Week 16 and Week 52 | Weeks 16 and Week 52
  GPPASI is common endpoints in clinical studies of GPP and is skin-based scoring systems. GPPASI is a modified composite index and an adaptation of the PASI score. The induration component has been substituted with a pustule component, with an overall score range from 0 (least severe) to 72 (most severe). Higher scores indicate more severe GPP. The five grades of severity for erythema, scaling, and pustulation correspond to 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. The score for each body region is calculated (the product of the sum of severity scores and its corresponding BSA score for erythema, scaling, and pustulation, multiplied by a weighting factor for each body region) and then the total GPPASI score determined (the sum of the individual scores from all body regions.
Change from Baseline in Japanese Dermatological Association Severity Index (JDASI) Score at Week 16 and Week 52 for Participants with Generalized Pustular Psoriasis | Week 16 and Week 52
  The Japanese Dermatological Association severity index (JDASI) assesses the systemic symptoms by laboratory changes. With the JDASI the skin is evaluated using three criteria (1) erythema area (overall), (2) erythema area with pustules and (3) oedema area. Scoring ranges from 3 to 0 (severe, moderate, mild, none) with a maximum of nine points. For systemic involvement pyrexia, white blood cell count, C reactive protein (CRP) and serum albumin with scores ranging from 2 to 0 (maximum 8 points) are assessed. The total JDASI score of GPP is the sum of both categories and categorizes as severe (17-11 points), moderate (10-7 points) or mild (0-6 points). Higher scores indicate more severe GPP.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (20):
- Japan (20):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Kimitsu Chuo Hospital, Kisarazu, Chiba
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu, Fukuoka
  - Isesaki Municipal Hospital, Isesaki, Gunma
  - Kobe University Hospital, Kobe, Hyōgo
  - Tokai University Hospital, Isehara, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Saitama Medical University Hospital, Iruma, Saitama
  - St.Luke's International Hospital, Chūō, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Fukuoka University Hospital, Fukuoka
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Okayama University Hospital, Okayama
  - Nippon Life Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/